CLINICAL TRIAL: NCT06501872
Title: Safety and Effectiveness of Physician-Modified Fenestrated and Branched Aortic Endografting for the Treatment of Thoracoabdominal and Pararenal Aortic Aneurysms
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bjoern D. Suckow (Other)
Responsible Party: Sponsor-Investigator, Bjoern D. Suckow, Associate Professor of Vascular Surgery, Dartmouth-Hitchcock Medical Center
Organization: Dartmouth-Hitchcock Medical Center (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY02002274
Record Dates: First submitted 2024-07-08; First posted 2024-07-15 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Aortic Aneurysm
Keywords: Aortic Aneurysm
MeSH Terms: conditions — Aortic Aneurysm

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Main Arm (Experimental): Use of a physician-modified fenestrated Cook Zenith Alpha Thoracic Endovascular Graft for the endovascular treatment of asymptomatic, non-ruptured thoracoabdominal aortic aneurysms of any Crawford extent (I-V) meeting traditional size criteria for open surgical repair.
  Interventions: Device: Physician-modified aortic endograft
- Expanded Access Arm (Experimental): Use of a physician-modified fenestrated Cook Zenith Alpha Thoracic Endovascular Graft for the endovascular treatment of asymptomatic, non-ruptured thoracoabdominal, thoracic, or abdominal aortic aneurysms of any Crawford extent (I-V) meeting traditional size criteria for open surgical repair in an expanded use population.
  Interventions: Device: Physician-modified aortic endograft

INTERVENTIONS:
Device: Physician-modified aortic endograft — Use of physician-modified fenestrated Cook Zenith Alpha Thoracic Endovascular Graft for the endovascular treatment of asymptomatic, non-ruptured thoracoabdominal aortic aneurysms of any Crawford extent (I-V) meeting traditional size criteria for open surgical repair.

SUMMARY:
The primary clinical objective of this study is to evaluate the safety and effectiveness of a physician-modified, fenestrated and branched aortic endoprosthesis for the treatment of thoracoabdominal aortic aneurysms (TAAAs). The goal of the primary analysis is to demonstrate both the safety and effectiveness of using a physician-modified fenestrated Cook Zenith Alpha Thoracic Endovascular Graft as compared to previously published results of open surgical replacement of the aneurysmal aorta.

DETAILED DESCRIPTION:
This study is a prospective, two-arm, traditional feasibility study of a physician modified fenestrated Cook Zenith Alpha Thoracic Endovascular Graft base device in adult patients meeting traditional size criteria for open surgical treatment of thoracoabdominal aortic aneurysms (TAAAs). Patients meriting surgical treatment of their aneurysm that also meet inclusion and exclusion criteria will be eligible for enrollment. Patients will be followed for 5 years post procedure.

ELIGIBILITY:
Main Arm Inclusion Criteria:

* Must be a man or woman 50 years of age or older by the date of informed consent
* Must have a thoracoabdominal aortic aneurysm of any Crawford classification (extent I-V) that extends no more proximal than the left subclavian artery.
* Must have an aneurysm size that meets standard indications for surgical repair (6.0 cm in maximum diameter in the descending thoracic aorta, or 5.5 cm in maximum diameter in the abdominal aorta)
* Must be considered, in the judgement of the Investigator, to be a high- risk candidate for open surgical repair
* Must commit to comply with the five-year study assessment schedule of events
* Must have a non-aneurysm-related life expectancy, in the judgement of the Investigator, of greater than 2 years

Expanded Selection Inclusion Criteria:

* Must be a man or woman 50 years of age or older by the date of informed consent
* Must have a thoracic, thoracoabdominal, or abdominal aortic aneurysm that necessitates coverage of one or more visceral vessels (celiac, superior mesenteric, or renals) for establishment of proximal and/or distal seal. The aneurysm must not extend proximal to the left subclavian artery, or, in the setting of more proximal disease, that disease must have been previously treated.
* Must have an aneurysm size that meets standard size indications for surgical repair (6.0 cm in maximum diameter in the descending thoracic aorta, or 5.5 cm in maximum diameter in the abdominal aorta); or, in the judgment of the Investigator, has aneurysm characteristics that portend a high risk of near-term rupture
* In the setting of an aortic dissection the following criteria must exist:

  * Access into the true lumen from the groin and at least one supra-aortic trunk vessel
  * A sealing zone in the target aorta (or surgical graft) that is proximal to the primary dissection, such that a stent graft would be anticipated to seal off the dissection lumen
  * A sealing zone in the target supra-aortic trunk vessels that is distal to the dissection, anticipated to seal off the dissection lumen, or surgically created
  * A true lumen size large enough to deploy the device and still gain access into the target branches
* Must be considered, in the judgement of the Investigator, to be a high-risk candidate for open surgical repair
* Patient must be able to provide informed consent
* Must commit to comply with the five-year study assessment schedule of events
* Must have a non-aneurysm-related life expectancy, in the judgement of the Investigator, of greater than 2 years

Main Arm Exclusion Criteria:

* Aneurysm due to acute or chronic dissection, intramural hematoma, penetrating aortic ulceration, pseudoaneurysm, mycotic aneurysm, or traumatic transection
* Ruptured or acutely symptomatic aortic aneurysm
* Known connective tissue disorder
* Imaging demonstrating any of the following:

  * Lack of 20 mm non-aneurysmal proximal seal zone (zone 3, or zone 2 with a carotid-subclavian bypass or transposition)
  * Lack of 15 mm non-aneurysmal distal seal zone(s) (aortic, common iliac, or external iliac)
  * Branch vessel target (renal, superior mesenteric, or celiac) < 5 mm or > 10 mm in average diameter
  * Untreated left subclavian artery stenosis or occlusion
  * Untreated unilateral or bilateral hypogastric artery occlusion
  * Signs that the inferior mesenteric artery is indispensable
  * Have branching, duplication, aneurysm, or untreatable stenosis of the celiac, superior mesenteric artery, or renal arteries that would preclude implantation of the investigational devices
* Known allergies to stainless steel, PTFE, polyester, polypropylene, nitinol, or gold
* History of anaphylaxis to contrast, with inability to prophylax appropriately.
* Have uncorrectable coagulopathy
* Have unstable angina
* Have a body habitus that would inhibit X-ray visualization of the aorta
* Have a major surgical or interventional procedure unrelated to the treatment of the aneurysm planned ≤30 days of the endovascular repair
* Known to be participating in any other clinical study which may affect performance of this - Ability to bear children
* Contraindication to oral antiplatelet therapy
* Prisoners or those on alternative sentencing
* Known systemic infection with potential for endovascular graft infection
* Anticipated need for MRI scanning within 3 months of insertion of investigational product
* Candidate for repair under the Instructions for Use of a commercially available, FDA-approved endovascular graft
* Can enroll in a manufacturer-sponsored clinical study at our institution or is willing and eligible to participate in a study with a manufacturer-made device at another institution.

Expanded Selection Exclusion Criteria:

* Known or suspected mycotic aneurysm
* Ruptured aneurysm with hemodynamic instability
* Known connective tissue disorder
* Imaging demonstrating any of the following:

  * Lack of 20 mm non-aneurysmal proximal seal zone (in either native aorta, elephant trunk graft, or aortic arch endograft)
  * Lack of 15 mm non-aneurysmal distal seal zone(s) (in either native aortoiliac vessels, prosthetic aortoiliac grafts, or aortoiliac endografts)
  * Branch vessel target (renal, superior mesenteric, or celiac) > 10 mm in average diameter
* Known allergies to stainless steel, PTFE, polyester, polypropylene, nitinol, or gold
* History of anaphylaxis to contrast, with inability to prophylax appropriately.
* Have uncorrectable coagulopathy
* Have a body habitus that would inhibit X-ray visualization of the aorta
* Have a major surgical or interventional procedure unrelated to the treatment of the aneurysm planned ≤ 30 days of the endovascular repair
* Known to be participating in any other clinical study which may affect performance of this device
* Ability to bear children
* Contraindication to oral antiplatelet therapy
* Prisoners or those on alternative sentencing
* Known systemic infection with potential for endovascular graft infection
* Anticipated need for MRI scanning within 3 months of insertion of investigational product
* Candidate for repair under the Instructions for Use of a commercially available, FDA- approved endovascular graft
* Can enroll in a manufacturer-sponsored clinical study at our institution or is willing and eligible to participate in a study with a manufacturer-made device at another institution
* Other conditions or comorbidities that, in the opinion of the Investigator, would exclude the patient

Ages: 50 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-12-10 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2031-09 (Estimated)

PRIMARY OUTCOMES:
30 day survival | 30 days
  Percent of patients who survive 30 days following surgery
Major Adverse Events (MAE) at 30 days following surgery | 30 days
  Percent of patients who development major adverse events at 30-days following surgery including the following:
  * All-cause mortality
  * Loss of major organ or system function
  * Renal failure necessitating hemodialysis
  * Small or large bowel ischemia necessitating surgical or endovascular intervention
  * Hepatic ischemia necessitating surgical or endovascular intervention
  * Gastric ischemia necessitating surgical or endovascular intervention
  * Paraparesis
  * Paraplegia
  * Stroke (Modified Rankin Score of 2 or greater)
  * Myocardial infarction
  * Ventilator dependence > 72 hours
  * Lower extremity ischemia necessitating surgical or endovascular intervention
  * Need for surgical or endovascular reintervention
Treatment success at 12 months following surgery | 12 months
  Percent of patients achieving treatment success through 1 year.
Technical success at 12 months following surgery | 12 months
  Technical success is assessed 12 months following surgery and is defined as a composite of: successful delivery, without need for unanticipated corrective intervention related to delivery; successful and accurate deployment at the intended implantation site; and successful withdrawal, without need for unanticipated correct intervention related to withdrawal.

SECONDARY OUTCOMES:
Technical success on the day of surgery | Day of Surgery
  Percent of patients achieving technical success on the day of surgery, defined as the composite of; successful delivery, successful and accurate deployment, successful withdrawal.
Aneurysm rupture | Day of Surgery
  Percent of patients developing aneurysm rupture
Conversion to open repair | Day of Surgery
  Percent of patients necessitating conversion to open repair. This is assessed intraoperatively. In case of a device deployment failure or intraoperative aneurysm rupture, emergent conversion to open repair via laparotomy, thoracotomy, or thoracoabdominal aortic exposure may become necessary. Patients undergoing such intraoperative conversion will be considered to have met this endpoint.
Access site complication (Femoral or Iliac) | Day of Surgery
  Percent of patients suffering access site complication (femoral or iliac). If femoral or iliac rupture occurs intraoperatively, or if femoral or iliac flow-limiting dissection or occlusion is identified intraoperatively or on the day of surgery, patients will be considered to have met this outcome.
Lower extremity ischemia | Day of Surgery
  Percent of patients developing lower extremity ischemia. This will be assess intraoperatively and on the day of surgery. If patients have lower extremity pulses either absent or diminished compared to baseline, with associated pain, sensory deficits or motor deficits on clinical evaluation, patients will be considered to have met this outcome.
Lower extremity compartment syndrome | Day of Surgery
  Percent of patients developing lower extremity compartment syndrome. In patients with lower extremity pain to passive motion post-operatively, invasive pressure measurement of the four calf compartments will be performed. If compartment pressures are greater than 30 in any compartment, patients will be considered to have met this outcome.
Stroke | Day of Surgery
  Percent of patients developing stroke - Modified Rankin Score (MRS) of 2 or greater). In patients with altered mental status or lateralizing motor or sensory deficits, MRI of the brain will be performed. If diffusion weighted MRI imaging demonstrates an intracranial lesion, a modified Rankin score will be calculated. If MRS is 2 or greater, patients will be considered to have met this outcome
Paraplegia | Day of Surgery
  Percent of patients developing paraplegia. Patients with complete absence of lower extremity motor function in one or both legs will be considered to have met this outcome.
Paraparesis | Day of Surgery
  Percent of patients developing paraparesis. Patients will undergo lower extremity motor strength assessment post-operatively on a standard 0 to 5 scale. If greater than 0 but less than 5 in either extremity, patients will be considered to have met this outcome.
Death during surgery | Day of Surgery
  Percent of patients who die during surgery
Survival rate | At 30, 183 days; 1, 2, 3, 4 and 5 years
  Percent of patients who survive
Major Adverse Events (MAEs) | At 30, 183 days; 1, 2, 3, 4 and 5 years
  Percent of patients that development MAEs
Treatment success | At 30, 183 days; 2, 3, 4 and 5 years
  Percent of patients achieving treatment success
Aneurysm-Specific Quality of Life Survey | At Screening, 30, 183 days; 2, 3, 4 and 5 years
  Assessment of quality of life using a validated disease-specific AAA survey. It will be measured using this survey.

CONTACTS AND LOCATIONS:
Overall Officials: Bjoern D Suckow, MD, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (1):
- Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire, United States

IPD SHARING:
Plan to Share IPD: No
No plan to share individual participant data (IPD) exists at this time.